CLINICAL TRIAL: NCT03827928
Title: The Acceptability, Feasibility, and Impact of a Group-based Yoga and Psychoeducation Program for Community-dwelling Adults With Multiple Sclerosis: A Randomized, Cross-over Pilot Study
Brief Title: LoveYourBrain Yoga for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Andrew D. Smith III, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D19058
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Fatigue; Anxiety; Depression
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga/meditation (Experimental): A 6-week yoga/meditation intervention.
  Interventions: Behavioral: Yoga/meditation
- Wait list (No Intervention): A wait list control period.

INTERVENTIONS:
Behavioral: Yoga/meditation — A 6-week yoga and meditation program with psychoeducation components, delivered through community-based yoga sessions. This program offers structured instruction: 10 minutes of breathing exercises to calm the nervous system, 45 minutes of gentle yoga to improve strength, flexibility, and balance, 15 minutes of guided meditation to enhance attention control, emotional regulation, and self-efficacy, and 20 minutes of facilitated discussion with psychoeducation to build community connection and skills in resilience.
  Arms: Yoga/meditation

SUMMARY:
The purpose of the study is to assess the feasibility of a 6-week yoga and meditation intervention for people with multiple sclerosis (MS). The study will evaluate the impact of the program on fatigue, anxiety, depression, positive affect, and other measures. A sub-study will collect brain images using MRI on 2 subjects before and after the intervention to identify potential biological markers of MS related-fatigue.

DETAILED DESCRIPTION:
This study will recruit 20 subjects with multiple sclerosis (MS) to participate in a 6-week yoga/meditation program. Subjects will be randomly assigned to one of two groups. The first group will complete the yoga/meditation classes, followed by a waiting period. The second group will go through a waiting period, followed by yoga/meditation classes. Two subjects assigned to classes during the first session will be selected to participate in an MRI sub-study to look for biomarkers of MS-associated fatigue. All subjects will complete questionnaires and assessments during 3 clinic visits - at baseline, in between the class sessions, and at the end of the study. Questionnaires will also be mailed to subjects 6 weeks after the last study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Sclerosis with EDSS score equal to or less than 6 (within last year)
2. 18 years of age or older
3. Ability to ambulate without assistance from a device or person
4. Subjects taking medications for depression, fatigue, or anxiety must be stable for 8 weeks prior to baseline
5. Able to read, write, and speak English
6. Willing to refrain from participating in yoga or meditation outside of the study for the duration of enrollment
7. Willing and able to give informed consent

Exclusion Criteria:

1. Participation in yoga and/or meditation more than twice within 8 weeks prior to baseline.
2. MS symptom exacerbation in the 8 weeks before baseline or other serious medical conditions that would impair ability to participate in the study.
3. Any other reason that, in the investigator's opinion, would exclude the subject from participation in the study.
4. Contraindication to scanning, including but not limited to ferromagnetic metal in the body, claustrophobia, inability to lie still or otherwise tolerate being in the scanner.
5. Pregnant women must be excluded from the imaging component of the study due to unknown but possible risk of fetal exposure to the scanner. Women of child-bearing potential will take a confidential pregnancy test immediately prior to each scan session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a yoga intervention study | At the clinic visit immediately following the yoga class session
  The feasibility will be determined by the completion rates of the intervention. If fewer than 50% of subjects complete the intervention, it will be deemed unfeasible in the current format.

SECONDARY OUTCOMES:
Change in subject self-rated fatigue | Through study completion, approximately 22 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue scale for MS: 8-item measure of fatigue. Scale range 8 to 40. A lower score represents a better outcome.
Change in subject self-rated self-efficacy | Through study completion, approximately 22 weeks
  Liverpool Self-efficacy scale: 17-item measure of self-efficacy. Scale range 17 to 68. A higher score represents a better outcome.
Change in subject self-rated anxiety | Through study completion, approximately 22 weeks
  Neuro-Quality of Life (QOL) v1.0 Anxiety - Short Form: 8-item measure of anxiety. Scale range 8 to 40. A lower score represents a better outcome.
Change in subject self-rated depression | Through study completion, approximately 22 weeks
  Neuro-Quality of Life (QOL) v1.0 Depression - Short Form: 8-item measure of depression. Scale range 8 to 40. A lower score represents a better outcome.
Change in subject self-rated positive affect | Through study completion, approximately 22 weeks
  Neuro-Quality of Life (QOL) v1.0 Positive affect and well-being - Short form: 9-item measure of positive affect and well-being. Scale range 8 to 48. A higher score represents a better outcome.
Change in subject cognition/processing speed | Through study completion, approximately 22 weeks
  Single Digit Modalities Test: Measure of cognition/processing speed. Score range 0 to 110. A higher score represents a better outcome.
Change in subject self-rated sleep disturbance | Through study completion, approximately 22 weeks
  Neuro-QOL v1.0 Sleep disturbance - Short Form: 8-item measure of sleep disturbance. Scale range 8 to 40. A lower score represents a better outcome.
Change in subject self-rated pain interference | Through study completion, approximately 22 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) v1.0 Pain Interference - Short Form 6b: 6-item measure of sleep disturbance. Scale range 6 to 30. A lower score represents a better outcome.
Change in subject self-rated quality of life | Through study completion, approximately 22 weeks
  Multiple Sclerosis Impact Scale (MSIS-29): 29-item measure of quality of life. Scale range 29 to 145. A lower score represents a better outcome.
Change in subject self-rated cognitive function | Through study completion, approximately 22 weeks
  Neuro-Quality of Life (QOL) v2.0 Cognitive Function - Short Form: 8-item measure of cognitive function. Scale range 8 to 48. A higher score represents a better outcome.
Satisfaction rating of 6-week yoga program on a scale of 1 - 10 | At the clinic visit immediately following the yoga/meditation class session
  Satisfaction scale: Subjects will rate their satisfaction with the yoga program on a scale of 1 - 10. Higher scores indicate a better rating.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No